CLINICAL TRIAL: NCT04598178
Title: Normative Data for the Quick Mild Cognitive Impairment-Taiwan Version (Qmci- TQ) in a Taiwanese Sample
Brief Title: Normative Data for the Qmci-TW in a Taiwanese Sample
Status: Completed | Type: Observational
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 202002051RINA
Record Dates: First submitted 2020-10-18; First posted 2020-10-22 (Actual); Last update posted 2021-05-06 (Actual); Status verified 2021-04

CONDITIONS: Postoperative Cognitive Dysfunction
MeSH Terms: conditions — Postoperative Cognitive Complications

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Taiwan Cohort: For normative Taiwan people, cognitive function will be assessed by the Taiwan version of questionnaire Qmci (Qmci-TW) on Day 0, Day 2, Day 180.

SUMMARY:
Many perioperative factors have been pointed out as the risk factors for postoperative cognitive dysfunction, which may occur immediately after the surgery, days after the surgery, or months after the surgery. Quick mild cognitive impairment screen (Qmci) is a sensitive and specific test to differentiate mild postoperative cognitive dysfunction. However, the learning effect have been raised as a bias when we repeated the same test for one person at different timing. Thus the study is designed to collected the Normative Data in series for the Qmci-TW in a Taiwanese Sample.

ELIGIBILITY:
Inclusion Criteria:

* adults no less than 20years old

Exclusion Criteria:

* pregnant women
* patients with respiratory failure [forced expiratory volume at one second (FEV1)/ forced vital capacity (FVC) < 70 % and FEV1 < 50%]
* patients with heart failure(NYHA score =III、IV)
* patients with chronic kidney disease (eGFR< 60 ml.min-1.1.73m-2)
* patients with liver failure
* patients with ongoing infection
* patients have surgery or hospital admission in the past half year

Min Age: 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Normative taiwan people
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2020-08-04 (Actual); Primary Completion 2021-02-27 (Actual); Study Completion 2021-02-27 (Actual)

PRIMARY OUTCOMES:
cognitive function by the Taiwan version of questionnaire Qmci (Qmci-TW) | 180 days
  Qmci is a screening assessment developed to detect mild cognitive impairment. It's a 100-point test administered in approximately 10 minutes. A score of 60 or over is considered to be normal. The validity of the Taiwan version of Qmci has been established.

CONTACTS AND LOCATIONS:
Overall Officials: Fon-Yih Tsuang, Ph.D., Principal Investigator — National Taiwan University Hospital
Locations (1):
- NTUH, Taipei, Taiwan, Taipei, Taiwan

REFERENCES:
- [Background] Steinmetz J, Christensen KB, Lund T, Lohse N, Rasmussen LS; ISPOCD Group. Long-term consequences of postoperative cognitive dysfunction. Anesthesiology. 2009 Mar;110(3):548-55. doi: 10.1097/ALN.0b013e318195b569. PMID 19225398
- [Background] Alam A, Hana Z, Jin Z, Suen KC, Ma D. Surgery, neuroinflammation and cognitive impairment. EBioMedicine. 2018 Nov;37:547-556. doi: 10.1016/j.ebiom.2018.10.021. Epub 2018 Oct 19. PMID 30348620
- [Background] Monk TG, Weldon BC, Garvan CW, Dede DE, van der Aa MT, Heilman KM, Gravenstein JS. Predictors of cognitive dysfunction after major noncardiac surgery. Anesthesiology. 2008 Jan;108(1):18-30. doi: 10.1097/01.anes.0000296071.19434.1e. PMID 18156878
- [Background] Lee MT, Chang WY, Jang Y. Psychometric and diagnostic properties of the Taiwan version of the Quick Mild Cognitive Impairment screen. PLoS One. 2018 Dec 3;13(12):e0207851. doi: 10.1371/journal.pone.0207851. eCollection 2018. PMID 30507928